CLINICAL TRIAL: NCT03289884
Title: Multi-metric Quantitative MRI for the Assessment of Hepatic Hydatid Disease- a Pilot Study
Brief Title: MR Assessment of Hepatic Hydatid Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 16/0811
Record Dates: First submitted 2017-08-07; First posted 2017-09-21 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Cystic Echincoccosis; Hydatid Disease
MeSH Terms: conditions — Echinococcosis | interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves; Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group (CE1): * All patients must have cystic lesions which must exceed 30mm in diameter.
  * All patients must be aged 16 or over and able to provide informed consent.
  * Patients will have an MRI scan (not involving ionising radiation)
  * Patients wil have an 'Ultrasound scan (not involving ionising radiation)'
  * Exclusion criteria include pregnancy and any contraindication to MRI (pacemaker, metallic implants, claustrophobia) and inability to give consent.
  Interventions: Other: MRI scan (not involving ionising radiation); Other: Ultrasound scan (not involving ionising radiation)
- CE group (CE2-4): * All patients must have hepatic CE, as confirmed by positive blood tests, with lesions identified on the standard of care MRI/CT scan, one or more of which must exceed 20 mm in diameter.
  * All patients must be aged 16 or over and able to provide informed consent.
  * All patients will have an MRI scan (not involving ionising radiation)
  * Patients wil have an 'Ultrasound scan (not involving ionising radiation)'
  * Exclusion criteria include pregnancy and any contraindication to MRI (pacemaker, metallic implants, claustrophobia) and inability to give consent.
  * Patients from the CE group undergoing surgery or aspiration will have fluid samples sent for analysis as part of standard clinical care. These cyst fluid samples will then be transported to the MRI scanner for Ex vivo scanning.
  Interventions: Other: MRI scan (not involving ionising radiation); Other: Ultrasound scan (not involving ionising radiation); Other: Ex vivo MRI scan of cyst fluid sample; Other: Aspiration of cyst fluid; Other: Blood test for confirmation of serum IgG levels consistent with hydatid infection

INTERVENTIONS:
Other: MRI scan (not involving ionising radiation) — The MRI study will be conducted by a trained MR radiographer, supervised by the nominated researcher
Other: Ultrasound scan (not involving ionising radiation) — The US scan will be conducted by a nominated researcher
Other: Ex vivo MRI scan of cyst fluid sample — The MRI study will be conducted by a trained MR radiographer, supervised by the nominated researcher
  Groups: CE group (CE2-4)
Other: Aspiration of cyst fluid — For patients undergoing surgery/radiologically guided aspiration the aspiration will be performed by a surgeon (at the Royal Free Hospital) or radiologist
  Groups: CE group (CE2-4)
Other: Blood test for confirmation of serum IgG levels consistent with hydatid infection — The blood sample will be drawn by a member of the clinical team
  Groups: CE group (CE2-4)

SUMMARY:
Hydatid disease is a major healthcare problem worldwide caused by infection that commonly affects the liver. Treatments for hydatid disease depend on how advanced the disease is and if the infection is active or not. Currently, doctors decide what stage the disease is at by looking at the appearance of liver on scans and by performing blood tests. It is however still very difficult to be certain if a treatment is working and when is the right moment to start and stop medication. Magnetic Resonance Imaging (MRI) scanning is a safe and non-invasive way of imaging the liver that can provide detailed information not just about what the liver looks like but also other information about the chemical composition of normal and diseased liver tissue. MRI is already widely used in the NHS for many liver conditions but it is unknown whether analysing the chemical composition will help decide on the stage and activity of hydatid liver disease. This study will allow comparison between MRI information about liver structure and composition with existing methods of assessing disease stage. If fluid is later obtained from the liver as part of usual clinical care (either using a needle with ultrasound or at the time of surgery), this study will also compare information about the fluid composition obtained from MRI scanning, with the results obtained when analysing the fluid in the lab. This will help to develop a more accurate way of non-invasively assessing hydatid disease in the liver, in the future.

DETAILED DESCRIPTION:
Cystic echincoccosis (CE), caused by infection with the dog tapeworm, is a major worldwide healthcare problem with increasing prevalence in the developed world. Approximately 75% of CE involves the liver, with treatments incurring significant cost and patient morbidity.

The key to CE treatment is correct identification of active infection but differentiation from sterile disease is highly problematic. Current treatment guidelines base activity assessment on morphological assessment with ultrasound (US), serology and light-microscopy of samples obtained at aspiration/surgery when available. Serology however can take many years to become negative even following successful treatment and US evaluation is subjective. Assessment of disease 'activity' is therefore a major challenge, particularly once patients are undergoing treatment. The lack of accurate tools to assess treatment response has undermined the development of management guidelines, particularly concerning the optimum length of chemotherapy treatment and indications for surgical/image-guided intervention.

Quantitative MR methods present a potential solution to this challenge. Magnetic Resonance Spectroscopy (MRS) has shown promising ex vivo results in detecting the biochemical "signature" of active infection in cyst fluid, but has yet to be applied clinically. Alternative approaches including T1 mapping, susceptibility mapping and Diffusion Weighted Imaging/Intra-voxel Incoherent Motion are also potentially useful, but have little supportive data to date.

Non-invasive biomarkers of CE activity are therefore essential to defining specific treatment endpoints, particularly in the context of chemotherapy. Multiple quantitative MR methods could be used to develop composite biomarkers for disease activity. Identifying a new quantitative radiological 'fingerprint' for each stage of the natural life-cycle of hepatic CE will enable improved diagnosis and therapeutic triage.

To date, in vivo liver quantitative MRI has not yet been applied to this cohort of patients, thus representing a novel application of this technology to address an important clinical question.

With this pilot study, the investigators aim to demonstrate the potential of quantitative MRI methods in the assessment of active/inactive hepatic CE.

ELIGIBILITY:
Inclusion Criteria for Control group:

* All patients must have cystic lesions which must exceed 30 mm in diameter.
* All patients must be fasted and avoid caffeinated fluids for at least 4 hours prior to the scan.
* All patients must be aged 16 or over and able to provide informed consent.

Inclusion Criteria for the CE group:

* All patients must have hepatic CE, as confirmed by positive serology, with lesions identified on teh standard of care MRI/CT scan, one or more of which must exceed 20 mm in diameter.
* All patients must be fasted and avoid caffeinated fluids for at least 4 hours prior to the scan.
* All patients must be aged 16 or over and able to provide informed consent.

Exclusion Criteria:

* Pregnancy
* Any contraindication to MRI (pacemakers, metallic implants, claustrophobia ect.)
* Inability to give consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment will take place at the hydatid liver disease multidisciplinary team meetings where patients are discussed and considered for inclusion. These patients can be recruited via outpatient consultation clinics.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2017-08-14 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is MR spectroscopy metabolite | 1 year
  This will be assessed on water ratio

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom

REFERENCES:
- [Background] Brunetti E, Garcia HH, Junghanss T; International CE Workshop in Lima, Peru, 2009. Cystic echinococcosis: chronic, complex, and still neglected. PLoS Negl Trop Dis. 2011 Jul;5(7):e1146. doi: 10.1371/journal.pntd.0001146. Epub 2011 Jul 26. No abstract available. PMID 21814584
- [Background] Budke CM, Deplazes P, Torgerson PR. Global socioeconomic impact of cystic echinococcosis. Emerg Infect Dis. 2006 Feb;12(2):296-303. doi: 10.3201/eid1202.050499. PMID 16494758
- [Background] Anand S, Rajagopalan S, Mohan R. Management of liver hydatid cysts - Current perspectives. Med J Armed Forces India. 2012 Jul;68(3):304-9. doi: 10.1016/j.mjafi.2012.04.010. PMID 24532894 (Retraction: PMID 30510356 Med J Armed Forces India. 2017 Jan;73(1):104)
- [Background] Benner C, Carabin H, Sanchez-Serrano LP, Budke CM, Carmena D. Analysis of the economic impact of cystic echinococcosis in Spain. Bull World Health Organ. 2010 Jan;88(1):49-57. doi: 10.2471/BLT.09.066795. PMID 20428353